CLINICAL TRIAL: NCT05978037
Title: An Open Label Phase I/IIa Clinical Trial to Assess the Safety, Immunogenicity and Efficacy of the Malaria Vaccine Candidate RH5.2-virus-like Particle (VLP) in Matrix-MTM, and to Compare the Safety and Immunogenicity of the Malaria Vaccine Candidates RH5.2-VLP in Matrix-MTM and RH5.1 Soluble Protein in Matrix-MTM Used in Various Regimens
Brief Title: A Study to Assess the Safety and Effectiveness of Two Experimental Malaria Vaccines
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIO-001
Record Dates: First submitted 2023-07-14; First posted 2023-08-07 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Malaria; Malaria,Falciparum; Parasitic Disease; Vector Borne Diseases; Infections
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Parasitic Diseases; Vector Borne Diseases; Infections | interventions — Matrix-M

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: 10 µg RH5.2-VLP with Months 0,1 and 2 regimen. (Active Comparator): This arm will receive monthly regimen of 3 doses of 10 µg of RH5.2-VLP with 50 µg Matrix-M .
  Interventions: Biological: RH5.1 and/or RH5.2-VLP with Matrix-M
- Group 2: 10 µg RH5.2-VLP with Months 0,1 and 6 regimen. (Active Comparator): This arm will receive 3 doses of 10 µg of RH5.2-VLP with 50 µg Matrix-M at Months 0, 1 and 6 (delayed regimen) and after Growth Inhibition Activity (GIA) immunogenicity review, will proceed to receive Controlled Human Malaria Infection (CHMI) 4 weeks after the last vaccination.
  Interventions: Biological: RH5.1 and/or RH5.2-VLP with Matrix-M
- Group 3: 10 µg or 2 µg RH5.2-VLP with Months 0,1 and 6 regimen. (Active Comparator): This arm will receive 2 doses of 10 µg of RH5.2-VLP with 50 µg Matrix-M at Months 0, 1 and 1 doses of 2 µg of RH5.2-VLP with 50 µg Matrix-M at Month 6 (delayed-fractional regimen).
  Interventions: Biological: RH5.1 and/or RH5.2-VLP with Matrix-M
- Group 4: 10 µg RH5.2-VLP or 2 µg RH5.1 with Months 0,1 and 6 regimen. (Active Comparator): This arm will receive 2 doses of 10 µg of RH5.2-VLP with 50 µg Matrix-M at Months 0, 1 and 1 doses of 2 µg of RH5.1 with 50 µg Matrix-M at Month 6 (delayed-fractional regimen, Prime with RH5.2-VLP then Boost with soluble RH5.1).
  Interventions: Biological: RH5.1 and/or RH5.2-VLP with Matrix-M
- Group 5: 10 µg or 2 µg RH5.1 with Months 0,1 and 6 regimen. (Active Comparator): This control arm will receive 2 doses of 10 µg of RH5.1 with 50 µg Matrix-M at Months 0, 1 and 1 doses of 2 µg of RH5.1 with 50 µg Matrix-M at Month 6 (delayed-fractional regimen with RH5.1).
  Interventions: Biological: RH5.1 and/or RH5.2-VLP with Matrix-M
- Group 6: CHMI control (No Intervention): This control arm will be infectivity controls, so will not receive any vaccinations.
  Group 6 will only be recruited after observation of meeting positive GIA target.

INTERVENTIONS:
Biological: RH5.1 and/or RH5.2-VLP with Matrix-M — The RH5.1 protein consists of the entire full-length ectodomain of the PfRH5 antigen (amino acids E26 - Q526) with the sequence based on the 3D7 clone of P. falciparum.
  The RH5.2 protein consists of the "stabilised" core region of PfRH5 antigen with SpyTag fused at the C-terminus. The RH5.2-SpyTag protein is conjugated to hepatitis B surface antigen (HBsAg)-SpyCatcher to produce the final RH5.2-VLP vaccine.
  The Matrix-M has been developed and manufactured by Novavax AB and is presented as a liquid solution in a glass vial.
  Arms: Group 1: 10 µg RH5.2-VLP with Months 0,1 and 2 regimen.; Group 2: 10 µg RH5.2-VLP with Months 0,1 and 6 regimen.; Group 3: 10 µg or 2 µg RH5.2-VLP with Months 0,1 and 6 regimen.; Group 4: 10 µg RH5.2-VLP or 2 µg RH5.1 with Months 0,1 and 6 regimen.; Group 5: 10 µg or 2 µg RH5.1 with Months 0,1 and 6 regimen.

SUMMARY:
Malaria is a major public health problem. There were around 240 million cases of malaria and 627,000 deaths worldwide in 2020. There is a great need for a safe, effective malaria vaccine and the team at University of Oxford is trying to make vaccine(s) which can prevent serious illness and death.

This study is being done to assess an experimental malaria vaccine for its ability to prevent malaria illness. This is done using a 'blood-stage challenge model'. This is when volunteers are infected with malaria parasites using malaria-infected red blood cells.

The vaccine we are testing in this part of the study is called "RH5.2-VLP". It is given with an adjuvant called "Matrix-M". This is a substance to improve the body's response to a vaccination. RH5.2-VLP is being tested for the first time in humans in this trial. The Matrix-M adjuvant has been given to tens of thousands of people, with no major concerns, such as illness.

The aim is to use this vaccine and adjuvant to help the body make an immune response against parts of the malaria parasite. This study will assess:

1. The safety of the vaccine in healthy participants.
2. The response of the human immune system to the vaccine.
3. The ability of the vaccine to prevent malaria illness (Group 2 only). We will do this by giving healthy adult participants (aged 18-45) three of the vaccines and/or expose participants to malaria infection at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital in Oxford. We will then do blood tests and collect information about any symptoms that occur after vaccination. There will be 19 to 54 visits, lasting between 3 months to 2 years and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy adult aged 18 to 45 years

  * Able and willing (in the Investigator's opinion) to comply with all study requirements.
  * Willing to allow the Investigators to discuss the volunteer's medical history with their GP
  * Participants of childbearing potential only: must practice continuous effective contraception for the duration of the study (see section 11.10)
  * Agreement to refrain from blood donation for the duration of the study
  * Able and willing to provide written informed consent to participate in the trial

Additional inclusion criteria for groups 2 and 6:

* Negative haemoglobinopathy screen (including sickle cell disease and alpha and beta thalassaemia) and normal G6PD levels
* Agreement to permanently refrain from blood donation, as per current UK Blood Transfusion and Tissue Transplantation Services guidelines (89)
* Reachable (24 hours a day) by mobile phone during the period between CHMI and completion of antimalarial treatment
* Willingness to take a curative anti-malaria regimen following CHMI
* Able to answer all questions on the informed consent questionnaire correctly at first or second attempt
* Able to travel to CCVTM without using public transport

Exclusion Criteria:

* • History of clinical malaria (any species) or previous participation in any malaria (vaccine) trial or CHMI

  * Travel to a clearly malaria endemic locality during the study period or within the preceding six months
  * Use of immunoglobulins or blood products (e.g. blood transfusion) in the last three months
  * Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days following each study vaccination, with the exception of COVID-19 and flu vaccines, which should not be received between 14 days before to 7 days after any study vaccination
  * Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period
  * Concurrent involvement in another clinical trial involving an investigational product or planned involvement during the study period
  * Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data, as assessed by the Investigator
  * Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
  * History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
  * Any history of anaphylaxis in relation to vaccinations
  * Pregnancy, lactation or intention to become pregnant during the study
  * History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
  * History of serious psychiatric condition that may affect participation in the study
  * Any other serious chronic illness requiring hospital specialist supervision
  * Suspected or known current alcohol misuse as defined by an alcohol intake of greater than 25 standard UK units every week
  * Suspected or known injecting drug use in the 5 years preceding enrolment
  * Hepatitis B surface antigen (HBsAg) detected in serum
  * Seropositive for hepatitis C virus (antibodies to HCV) at screening (unless volunteer has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV ribonucleic acid (RNA) PCR at screening for this study)
  * Volunteers unable to be closely followed for social, geographic or psychological reasons.
  * Any clinically significant abnormal finding on biochemistry or haematology blood tests or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested.
  * Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
  * Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Additional exclusion criteria for Groups 2 and 6:

* Body weight <50 kg or Body Mass Index (BMI) <18.0 at screening
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin)
* Use of anti-malarials within 30 days of CHMI
* Receipt of a COVID-19 vaccine within 2 weeks before the day of CHMI or planned receipt of a COVID-19 vaccine or prior to expected completion of antimalarial treatment (around 2 to 3 weeks after day of challenge based on experience in previous P. falciparum CHMI studies to date)
* An estimated ten-year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE).
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone
* Any other contraindications/known hypersensitivities to both Riamet and Malarone
* Any clinical condition known to prolong the QT interval
* History, or evidence at screening, of clinically significant arrhythmias, including clinically relevant bradycardia, prolonged QT interval or other clinically relevant ECG abnormalities
* Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia
* Family history of congenital QT prolongation or sudden death
* Positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease
* History of sickle cell anaemia, sickle cell trait, thalassaemia or thalassaemia trait, G6PD deficiency or any haematological condition that could affect susceptibility to malaria infection

Additional exclusion criteria for optional FNA in Groups 1 and 3:

* Regular use of anticoagulation or antiplatelet medication likely to induce bruising or bleeding on fine needle aspiration.
* Any confirmed or suspected bleeding disorders.
* History of lymphatic disorders (e.g. lymphoedema).
* History of allergic disease or reactions to local anaesthetic such as lidocaine.
* Any history of anaphylaxis in relation to local anaesthetic such as lidocaine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of RH5.2-VLP and RH5.1 in Matrix-M in healthy volunteers at different doses and used in various regimens by assessing the occurrence of solicited local reactogenicity signs and symptoms | 7 days following each vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following each vaccination. These will be tabulated, detailing frequency, duration and severity of AEs. Haematological and biochemical laboratory values will be presented according to local grading scales.
To assess efficacy of RH5.2-VLP in Matrix-M by assessing its impact on parasite multiplication rate (PMR) in vaccinated volunteers compared to infectivity controls, against P. falciparum in a blood-stage controlled human malaria infection (CHMI) model. | Maximum 21 days following CHMI
  Comparison of the PMR of the volunteers in Group 2 to the PMR of the malaria naive controls (Group 6) over 21 days of follow up period post-CHMI. PMR values will be collected initially as quantitative PCR data and calculated using a mathematical modelling.

SECONDARY OUTCOMES:
To assess the humoral immunogenicity of RH5.2-VLP with Matrix-MTM and RH5.1 soluble protein with Matrix-M when administered to healthy volunteers at different doses and used in various regimens, with comparison before and after vaccination | From a number of key timepoints (Baseline up to day 790 (dependant on group))
  Serum ELISA response, antigen-specific antibody avidity measurement, antigen-specific antibody subclass/isotype measurement, quantitative antigen-specific IgG antibody levels (µg/mL readout) over time - analysis of peak responses and longevity, with comparison before and after vaccination
To compare the anti-RH5 serum IgG functional immunogenicity between the RH5.2-VLP and soluble RH5.1 protein when used at different doses and in various regimens | From a number of key timepoints (Baseline up to day 790 (dependant on group))
  In vitro GIA against 3D7 clone P. falciparum parasites using purified total IgG and a single-cycle pLDH readout assay, with comparison before and after vaccination.
To determine the phenotype of vaccine specific immune cells in axillary lymph nodes | Day 140 (group 1) and Day 266 (group 3)
  BCR sequencing with vaccine-specific B cells obtained from axillary lymph nodes to characterise the B cell repertoire (Group 1 & 3 only)
To determine the frequency of vaccine specific immune cells in axillary lymph nodes | Day 140 (group 1) and Day 266 (group 3)
  BCR sequencing with vaccine-specific B cells obtained from axillary lymph nodes to characterise the B cell repertoire (Group 1 & 3 only)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Minassian, Dr, Principal Investigator — angela.minassian@bioch.ox.ac.uk
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom